CLINICAL TRIAL: NCT04623411
Title: The Effect of Serious Game Simulation on Newborn Resuscitation Education of Nursing Students
Brief Title: Use of Serious Game Simulation on Newborn Resuscitation Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Sureyya Sarvan, PhD, Principal Investigator, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5154
Record Dates: First submitted 2020-11-04; First posted 2020-11-10 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Newborn; Vitality
Keywords: Newborn Resuscitation; Simulation; Serious game; Nursing Student
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This was pretest-posttest design, randomized controlled trial.
Who Masked: Participant
Masking Description: The control and intervention group will be formed by randomization. The intervention and control group will be defined as group 1 and group 2 for statistical analysis. Data analysis will be evaluated and reported by the statistician. Also the statistician will be blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Neonatal resuscitation training with classical method and serious game simulation method
  Interventions: Behavioral: Neonatal resuscitation training with classical method and serious game simulation method
- Control Group (Experimental): Neonatal resuscitation training with classical method.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Neonatal resuscitation training with classical method and serious game simulation method — After the theoretical training, the participants will be given technical information on the use of web-based neonatal resuscitation serious game simulation method.
  Each participant will be asked to apply this method at least three times.
  Arms: Intervention Group
Behavioral: Control Group — Neonatal resuscitation training with classical method
  Arms: Control Group

SUMMARY:
Neonatal death is one of the important indicators showing the development level of countries. Many newborn deaths are preventable. Preventable neonatal deaths arise from events such as birth asphyxia at the time of delivery. Nursing students receive neonatal resuscitation training with classical training methods and graduate without the opportunity to experience it in a clinical setting. The aim of the study is to evaluate the effectiveness of web-based serious game simulation method in neonatal resuscitation training given to nursing students.

DETAILED DESCRIPTION:
The study was planned as a randomized controlled trial with a single blind, pretest-posttest design. This study will be conducted in the Fall Semester of the 2020-2021 Academic Year with nursing students studying in the 3rd grade of Akdeniz University Faculty of Nursing between October and December 2020. An intervention and control group (intervention group: 50, control group: 50) will be formed from 100 students who accepted to participate in the study. Participants will be randomly allocated to one of the two groups. Pre-test and post-test will be applied to both groups before and after the training. Neonatal resuscitation training will be given online to the intervention and control group. After the theoretical training, web-based neonatal resuscitation serious game simulation will be applied to the intervention group. Ethics Committee and Institutional Permission was obtained for the study. In addition, written consent will be obtained from the participants. Statistical analysis will be done using SPSS 23.0 and significance will be evaluated at p <0.05. Support will be received in the analysis phase of the Statistical Information Unit of Akdeniz Universit It is predicted that the new information obtained from the data of the research will guide the methods used in education and new researches.

ELIGIBILITY:
Inclusion Criteria:

* Students who are volunteers, Those who attend the Neonatal Nursing Course, Nursing students in the 3rd grade, Students with laptops

Exclusion Criteria:

* Those with neonatal resuscitation certificate, Students without internet access

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-11-29 (Actual); Study Completion 2021-03-09 (Actual)

PRIMARY OUTCOMES:
Neonatal resuscitation knowledge level assessment questionnaire | Immediately before training and one week after training completion
  This 15-item multiple-choice questionnaire was developed by the researchers to evaluate the knowledge level of the participants. Each question will be evaluated as correct answer = 1 point, wrong answer = 0 points. Participants will fill in online before and after the training.
Evaluation of Newborn Resuscitation Practice Skills | Immediately before training and one week after training completion
  Serious game simulation software will be used to Assess Newborn Resuscitation Practice Skill. Participants will be expected to practice web-based neonatal resuscitation with serious game simulation and their skills will be evaluated. Each correct practice will be evaluated as sufficient 1 point and incorrect practice will be evaluated as 0 points.

SECONDARY OUTCOMES:
Student Satisfaction and Self-Confidence in Learning Scale | One week after training completion
  The scale consists of two sub-dimensions, "satisfaction with learning" and "self-confidence", in five-point Likert type, and a total of 13 items. There are five items in the satisfaction with learning sub-dimension and eight items in the self-confidence sub-dimension. Internal consistency coefficient of the scale: 0,90 The internal consistency coefficient of student satisfaction is 0.89, and the self-confidence in learning sub-dimension is 0.83.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Konyaaltı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wyckoff MH, Aziz K, Escobedo MB, Kapadia VS, Kattwinkel J, Perlman JM, Simon WM, Weiner GM, Zaichkin JG. Part 13: Neonatal Resuscitation: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S543-60. doi: 10.1161/CIR.0000000000000267. No abstract available. PMID 26473001
- [Result] Ghoman SK, Cutumisu M, Schmolzer GM. Simulation-Based Summative Assessment of Neonatal Resuscitation Providers Using the RETAIN Serious Board Game-A Pilot Study. Front Pediatr. 2020 Jan 31;8:14. doi: 10.3389/fped.2020.00014. eCollection 2020. PMID 32083041